CLINICAL TRIAL: NCT03806257
Title: Patient Mobility and Outcomes After Cardiac Surgery: a Randomized Controlled Trial
Brief Title: Patient Mobility and Outcomes After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sreekanth Cheruku, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 012018-090
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective design involving two study groups: 1) standard-of-care for cardiac physical therapy, and 2) enhanced protocol for cardiac physical therapy. Primary aim is to assess difference, if any, between groups for ICU and hospital length of stay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Subjects in the control arm will receive standard of care, which consists of mobilization to a bedside chair at least once, and ambulate one-half ICU circumference on postoperative day one. On postoperative days two through five, the subject will be mobilized to the bedside chair at least once, and ambulated at least once with target of one full ICU circumference. These subjects will receive gait training and safe ambulation education, and wear a FitBit Charge 2 watch for five days after surgery.
- Enhanced Physical Therapy Protocol (Experimental): Subjects in the experimental arm will recieve a FitBit Charge 2 watch, and will be mobilized to the bedside chair on postoperative day zero. On postoperative day two subjects will be mobilized to the bedside chair twice, ambulate one-half of the ICU circumference, and receive gait and safe ambulation training. On postoperative days two through five, subjects will mobilize to the bedside chair three times, and will be encouraged to ambulate three times, each time with a target of one full ICU circumference.
  Interventions: Other: Enhanced Physical Therapy Protocol

INTERVENTIONS:
Other: Enhanced Physical Therapy Protocol — A structured physical therapy protocol that requires subject to ambulate more frequently than the standard-of-care patient.
  Arms: Enhanced Physical Therapy Protocol

SUMMARY:
Standards for post-cardiac surgery physical interventions vary between insitutions and there are no published guidelines for national organizations in the U.S. The increasing body of evidence for the effectiveness of physical interventions coupled with variability in how these interventions are implemented suggests a critical need to prospectively determine the impact of clearly defined postoperative physical interventions. This randomized, controlled study seeks to determine the effectiveness of a three-pronged, enhanced, post-operative physical therapy protocol which includes 1) early mobilization, 2) frequent mobilization and ambulation, and 3) patient education on the outcomes of hospital lengths of stay and discharge disposition. The investigators will enroll 220 adult subjects undergoing elective CABG, mitral valve repair or replacement surgery, aortic valve surgery, or combined CABG/valve procedures. Subjects will be randomized to either the control (standard-of-care) group or intervention group (enhanced protocol), and followed for five days. Subjects in each group will wear a FitBit Charge 2 for the duration of the five days following surgery. This will provide both sleep activity and steps data that will be analyzed for sleep quality and distance walked. The primary aim is to assess the difference between groups for ICU and hospital length of stay.

DETAILED DESCRIPTION:
Patients will be identified based on pre-screening the cardiothoracic surgery schedule. Study staff will visit potential study subjects in the pre-surgical testing clinic to discuss the study's objectives and to ascertain subjects' interest in participating in the study. After providing informed consent, subjects will be randomized using SAS into either the interventional group or standard care group after their surgical procedure is complete and the subject has been transferred to the CVICU. After completion of the surgical procedure, patients who had a major perioperative complication such as stroke, myocardial infarction, pulmonary embolism, hemorrhage requiring massive transfusion (>10 units of PRBCs), intraoperative cardiac arrest, or intraoperative pulmonary arrest, will be considered screen failures and will not be randomized, since the investigators consider the patient enrolled once randomized. Patients randomized to the interventional group will undergo the enhanced physical therapy protocol which includes mobilization from bed to chair on the day of surgery and more frequent ambulation on the subsequent five days.

The main differences between the standard therapy (control) group and intervention group is the timing of post-operative mobilization and ambulation, as well as the point at which they receive gait and safe ambulation training. In the standard therapy group, the patients will receive a FitBit2 after their arrival on the ICU, withstanding any postoperative complications. On POD 1 the subjects routinely get up to the bedside chair with the help of an ICU nurse or physical therapist. The subjects will generally ambulate one-half the circumference of the ICU with assistance, though this is not enforced. On POD2 and onward, the standard therapy group typically will get up to the bedside chair at least once, as well as walk one-half circumference of the ICU, and will receive the standard physical therapy gait and ambulation training. The intervention group will have the FitBit2 watch placed on their wrist on POD 0, along with getting up to the bedside chair. On POD 1, the subjects will get up to the bedside chair twice (as tolerated by patient), and will be asked to walk one-half the ICU circumference. Additionally, the patient's physical therapy and gait/ambulation training will commence on POD 1. On POD 2, the subjects will get up to the bedside chair three times, and will be asked to attempt three walks with the goal of one full ICU circumference.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older undergoing scheduled, elective coronary artery bypass graft (CABG) surgery, mitral valve repair or replacement surgery, aortic valve repair or replacement surgery and combined CABG with one or more valve repair or replacement surgery.

Exclusion Criteria:

* Those who do not med the inclusion criteria
* Pregnant women
* Prisoners
* Those patients with skin or systemic infections
* Those patients who are paraplegic or quadriplegic
* Those patients who have allergies to polyurethane
* Any patient who experiences perioperative complications (e.g., stroke, myocardial infarction, pulmonary embolism, hemorrhage requiring massive transfusion (>10 units of PRBCs), intraoperative cardiac arrest, or intraoperative pulmonary arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Shorter ICU Length of Stay | 1.2 days
  Decrease days in ICU from average standard-of-care patient
Shorter Hospital Length of Stay | 2 days
  Decrease days in hospital from average standard-of-care patient

SECONDARY OUTCOMES:
Composite Clinical Outcome | 5 days
  Combined incidence of pulmonary atelectasis, pneumonia, venous thromboembolism, pulmonary embolism, and mortality.
Longer sleep duration with fewer awakenings | 8 hours sleep, less than 3 awakenings
  Sleep time that is longer than average standard-of-care patient

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We will not share data with any outside entity or non-IRB-approved personnel.

REFERENCES:
- [Background] Herdy AH, Marcchi PL, Vila A, Tavares C, Collaco J, Niebauer J, Ribeiro JP. Pre- and postoperative cardiopulmonary rehabilitation in hospitalized patients undergoing coronary artery bypass surgery: a randomized controlled trial. Am J Phys Med Rehabil. 2008 Sep;87(9):714-9. doi: 10.1097/PHM.0b013e3181839152. PMID 18716482